CLINICAL TRIAL: NCT04092231
Title: Subjective and Functional Outcome Measures to Evaluate Performance of Pediatric Cochlear Implant
Brief Title: Outcomes of Cochlear Implantation in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Amira Mohmed Ahmed Bakr (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Amira Mohmed Ahmed Bakr, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 1815
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Hearing Impaired Children
Keywords: Hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Thirty children were between two and five years of age at the time of implantation. All were congenital pre-linguistically bilateral profound sensorineural hearing loss. Reports about basic audiological evaluation which included air and bone conduction thresholds, speech audiometry for all the study group before the implantation were obtained. They had limited benefit from consistent use of hearing aid amplification and enrolled in a rehabilitation program focused on oral communication. they underwent unilateral CI with CI experience ranged from 6 months and above.
  Interventions: Behavioral: Early speech perception test

INTERVENTIONS:
Behavioral: Early speech perception test — The early speech test is one of the closed-set response speech discrimination tests,using object identification technique.It was carefully designed for estimation of speech perception abilities in very young children who have extremely low verbal abilities
  Other Names: Meaningful Auditory Integration Scale

SUMMARY:
The cochlear implant (CI) is the most important progress in the treatment for adults and children with severe to profound bilateral sensorineural hearing loss who do not receive adequa¬te benefit from hearing aids and making possible better results in auditory, linguistic, social and academic development.

DETAILED DESCRIPTION:
Tomblin JB et al.1997, Svirsky MA, 2004 reported that the early restoration of auditory ability by cochlear implants significantly improve the commu¬nication skills, albeit with varied results. Thoutenhoofd E 2005 concluded that while most children with cochlear implants become able to attend school regularly, other remain with significantly limited verbal communication skills

Earlier implantation for children with a congenital profound hearing loss appeared to provide improved potential for developing speech perception. which improved steadily with implant experience.

The speech perception can be defined as the process of imposing a meaningful perceptual experience from meaningless speech input, wich may be thought of involving a number of components as: detection, discrimination, identification, attention, memory and closure .

In the field of aural rehabilitation, speech perception assessment has an important and a critical role to select the signal processing strategy, to adjust the signal processor and to determine if appropriate benefit has been achived .

Young children,being considered apart of the language limited,difficult-to test population, efforts were directed towards construction of special hearing test to suit their reduced verbal language(Mc Lauchlin,1980).

The early speech test(EST) is one of these tests,which use low -verbal materials.

The early speech test is one of the closed-set response speech discrimination tests,using object identification technique.It was carefully designed for estimation of speech perception abilities in very young children who have extremely low verbal abilities.

Most studies on the impact of cochlear implants have focused on clinical assessments of efficacy (hearing and speech skills, and auditory thresholds). It is not clear how much clinical measures of efficacy (speech, hearing, and language measures) truly show the effectiveness of cochlear implants in general contexts (such as performance at home, at school, and in social settings). Vidas S et al 1992 reported that there is evidence that clinical assessment results do not correlate with performance in unstructured settings, these measures are only part for assessments of cochlear implant efficacy.

There are questionnaires that investigate the expectations of parents (Thoutenhoofd E 2005, Vaccari C, Marschark M. 1997, Spilker B, Revicki D.1996) their satisfaction level with implant, the stresses in this process8, and cochlear implant user and family quality of life .

* The Meaningful Use of Speech Scale (MUSS) questionnaire was used to analyze and measure speech skills (Nascimento et al 1997)and allows the examiner to evaluate a child skills in meaningful real world situation.

ELIGIBILITY:
Inclusion Criteria: Between 2 and 5 years of age at time of implantation

* Profound bilateral sensorineural hearing loss
* Arabic as the primary language in the home
* Realistic expectations of guardians
* Child must be enrolled in a post-operative rehabilitative/educational program that supports the use of cochlear implants and the development of auditory-based skills
* Willing and available to comply with all scheduled procedures as defined in the protocol
* Profound bilateral sensorineural hearing loss with average thresholds between ears of 90 dB HL or greater at 1000 Hz and aboveBehavioral test measures must include unaided threshold measures for the right and left ears using insert earphones; left-alone and right-alone aided sound field threshold measurements; and aided and unaided speech-awareness / detection thresholds (for each ear individually)
* Children accepted into the study must be able to demonstrate a consistent response to sound. If a child has no measurable hearing, he/she must be able to demonstrate a consistent response to vibrotactile stimuli.
* All children must have completed an appropriate trial period with optimally fit amplification prior to inclusion in the study.

Exclusion Criteria:Subjects with mental retardation (MR), below average mentality or any subject with behavioral problems, traumatic brain injury, additional significant disabilities (e.g., blindness, autism) or with auditory neuropathy were excluded from the study

-

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thirty children were between two and five years of age at the time of implantation. All were congenital pre-linguistically bilateral profound sensorineural hearing loss. Reports about basic audiological evaluation which included air and bone conduction thresholds, speech audiometry for all the study group before the implantation were obtained. They had limited benefit from consistent use of hearing aid amplification and enrolled in a rehabilitation program focused on oral communication. they underwent unilateral CI with CI experience ranged from 6 months and above.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
change in percent correct in speech perception as measured with single words presented in a closed set | 1 year
  ):-Change in percent correct in speech perception as measured with single words presented in a closed set. [ Time Frame: Speech perception will be compared baseline to 3 month post implant, baseline to 6 month post implant, baseline to 9 month post implant, baseline to 12 months post implant, baseline to 18 months post implant and baseline to 24 months post implant Closed set word identification presented by direct input to the speech processor using the Early Speech Perception (ESP)Test (Moog & Geers,1990), which is a test commonly used to assess young children with hearing loss 2-patient related benefits - improvements in hearing ability assessed via Meaningful Auditory Integration Scale.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavicchiolo S, Mozzanica F, Guerzoni L, Murri A, Dall'Ora I, Ambrogi F, Barozzi S, Cuda D, Schindler A. Early prelingual auditory development in Italian infants and toddlers analysed through the Italian version of the Infant-Toddler Meaningful Auditory Integration Scale (IT-MAIS). Eur Arch Otorhinolaryngol. 2018 Feb;275(2):615-622. doi: 10.1007/s00405-017-4847-6. Epub 2017 Dec 16. PMID 29248951
- [Background] Nilakantan A, Raj P, Saini S, Mittal R. Early Speech Perception Test Outcome in Children with Severe Sensorineural Hearing Loss with Unilateral Cochlear Implants Alone versus Bimodal Stimulation. Indian J Otolaryngol Head Neck Surg. 2018 Sep;70(3):398-404. doi: 10.1007/s12070-018-1398-0. Epub 2018 May 14. PMID 30211097
- [Background] Thomas E, El-Kashlan H, Zwolan TA. Children with cochlear implants who live in monolingual and bilingual homes. Otol Neurotol. 2008 Feb;29(2):230-4. doi: 10.1097/mao.0b013e31815f668b. PMID 18223450